CLINICAL TRIAL: NCT02870491
Title: Working With Community Health Workers to Increase Oral Rehydration Salt and Zinc Use to Treat Child Diarrhea in Uganda: A Cluster Randomized Controlled Trial
Brief Title: Working With Community Health Workers to Increase ORS Use in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: ZW-03-28-1983
Record Dates: First submitted 2016-08-09; First posted 2016-08-17 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Infantile Diarrhea; Diarrhea; Dehydration
Keywords: Child Diarrhea; Cluster Randomized Controlled Trial; Oral Rehydration; ORS; Zinc; Brac; Community Health Workers; Uganda
MeSH Terms: conditions — Diarrhea, Infantile; Diarrhea; Dehydration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (No Intervention): Existing standard of care.
- Free Distribute+Preemptive Delivery (Experimental): Community health workers (CHWs) will deliver oral rehydration salts (ORS) and zinc for free to all households in their catchment area with a child under 5-years-old at the beginning of the study.
  Interventions: Behavioral: Free Distribution; Behavioral: Preemptive Delivery
- Cost Sharing + Preemptive Delivery (Experimental): CHWs will visit all households with a child under 5-years-old at the beginning of the study and offer to sell ORS and zinc to caretakers at the time of the visit for them to store in their homes.
  Interventions: Behavioral: Preemptive Delivery
- Free Distribution Upon Retrieval (Experimental): CHWs will visit all households with a child under 5-years-old at the beginning of the study and inform caretakers that they have ORS and zinc available for free that caretakers can retrieved from the CHWs home if needed.
  Interventions: Behavioral: Free Distribution

INTERVENTIONS:
Behavioral: Free Distribution — Caretakers of children under 5-years-old will have access to free ORS and zinc
  Arms: Free Distribute+Preemptive Delivery; Free Distribution Upon Retrieval
Behavioral: Preemptive Delivery — Caretakers of children under 5-years-old will have ORS and zinc delivered to their home
  Arms: Cost Sharing + Preemptive Delivery; Free Distribute+Preemptive Delivery

SUMMARY:
The purpose of this study is to assess how free distribution and preemptive home delivery of oral rehydration salts (ORS) by community health workers affects ORS use. The investigators will measure the impact of the combination of the two interventions (free distribution + pre-emptive home delivery) as well as the impact of each intervention separately (free distribution without home delivery and pre-emptive home delivery without free distribution).

DETAILED DESCRIPTION:
This research aims to test the impact of a novel preemptive home-delivery intervention aimed at increasing the use of oral rehydration salts (ORS) and zinc for child diarrhea in Uganda. The intervention aims to increase availability of ORS and zinc and reduce barriers to access by having community health workers (CHWs) deliver the products directly to households for free prior to a diarrhea episode. Under this set-up, the products will be readily available for free immediately after a child comes down with diarrhea. Moreover, the investigators will disentangle the mechanisms through which the intervention could change product use by using a multi-armed approach that tests for the impact of free distribution and preemptive home-delivery separately (i.e. preemptive delivery but not free and free but not preemptive delivery). The investigators will use a four-arm cluster randomized controlled trial designed to measure the impact of each of the three interventions on ORS and zinc use for treating child diarrhea relative to a control group. The investigators will enroll 120 CHWs (each located in a different village) and randomly assign each to 1 of 4 groups:

Group 1 - Control: No intervention will take place. Caretakers will have standard access to ORS and zinc at local health facilities and pharmacies. Some CHWs in control villages could make household visits, however offers to sell diarrhea treatment preemptively are rare and CHWs are generally not the source of diarrhea treatment.

Group 2 - Household Visit + Free Distribution + Preemptive Delivery: CHWs will be provided a small incentive to visit all of the households in their catchment area that contain a child under 5-years-old (roughly 100 households) at the beginning of the study. CHWs will train caretakers on the dangers of diarrhea and the importance of ORS and zinc use. CHWs will then offer to give ORS and zinc to caretakers for free to store in their homes.

Group 3 - Household Visit + Cost Sharing + Preemptive Delivery: CHWs will be provided a small incentive to visit all of the households in their catchment area that contain a child under 5-years-old at the beginning of the study. CHWs will train caretakers on the dangers of diarrhea and the importance of ORS and zinc use. CHWs will then offer to sell ORS and zinc to caretakers at their standard subsidized price (roughly USD$0.40 in total per treatment course) to store in their homes.

Group 4 - Household Visit + Free Distribution Upon Retrieval: CHWs will be provided a small incentive to visit all of the households in their catchment area that contain a child under 5-years-old at the beginning of the study. CHWs will train caretakers on the dangers of diarrhea and the importance of ORS and zinc use. CHWs will then inform caretakers that they have ORS and zinc available for free that caretakers can retrieved from the CHWs home if needed. The average distance to the CHWs household is about 15 minutes.

Groups 2-4 compared to Group 1 measures the impact of each of the different ways of arranging the program. Group 3 compared to Group 2 measures the price effect. Group 4 compared to Group 2 measures the distance/convenience effect. Group 2 compared to Group 1 measures the combination of the price and distance/convenience effect.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-59 months that reside on a village recruited to participate in the study will be included in the intervention. Only children with a diarrhea episode 4-weeks prior to data collection will be included in the analysis.

Exclusion Criteria:

* Children without a diarrhea episode in the weeks prior to data collection will be excluded from the analysis.

Max Age: 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7949 (Actual)
Dates: Start 2016-08; Primary Completion 2017-06 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Oral rehydration salt (ORS) use | Last 4 weeks
  Caretaker-reported ORS use to treat a diarrhea episode in the last 4 weeks

SECONDARY OUTCOMES:
Oral rehydration salt (ORS) with Zinc use | Last 4 weeks
  Caretaker-reported ORS + zinc use to treat a diarrhea episode in the last 4 weeks
Antibiotic use | Last 4 weeks
  Caretaker-reported antibiotic use to treat a diarrhea episode in the last 4 weeks
Time to Oral rehydration salt (ORS) use | Last 4 weeks
  Caretaker-reported time from diarrhea initiation to ORS use
Time to zinc use | Last 4 weeks
  Caretaker-reported time from diarrhea initiation to zinc use

OTHER OUTCOMES:
Oral rehydration salt (ORS) use | Last 7 days
  Caretaker-reported ORS use to treat a diarrhea episode in the last 7 days
Oral rehydration salt (ORS) use | current diarrhea episode up to 4 weeks
  Caretaker-reported ORS use to treat a current diarrhea episode

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to the public after the results are published